CLINICAL TRIAL: NCT01980667
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination With Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Study of Lurbinectedin (PM01183) in Combination With Cisplatin in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-008-13
Record Dates: First submitted 2013-10-22; First posted 2013-11-11 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Solid Tumors
Keywords: lurbinectedin; PM01183; tumors; cancer; Pharma Mar
MeSH Terms: conditions — Neoplasms | interventions — PM 01183; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lurbinectedin (PM01183) / cisplatin (Experimental): Patients will receive cisplatin as a 90-min i.v. infusion. In addition, patients will receive PM01183 as an i.v. infusion over 1-hour.
  Interventions: Drug: lurbinectedin (PM01183); Drug: Cisplatin

INTERVENTIONS:
Drug: lurbinectedin (PM01183) — lurbinectedin (PM01183) is presented as powder for concentrate for solution for infusion with two strengths, 1-mg and 4-mg vials.
Drug: Cisplatin — vials containing 1 mg/ml concentrate for solution for infusion

SUMMARY:
Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination with Cisplatin in Patients with Advanced Solid Tumors to determine the recommended dose (RD) of PM01183 in combination with cisplatin, to characterize the safety profile, the pharmacokinetics (PK) of this combination, to obtain preliminary information on the clinical antitumor activity and to conduct an exploratory pharmacogenomic (PGx) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent
* Age ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 1.
* Life expectancy ≥ 3 months.
* Patients with confirmed diagnosis of advanced solid tumors.
* Patients may have received ≤ 2 chemotherapy-containing lines in the advanced setting.
* Adequate bone marrow, renal, hepatic, and metabolic function (assessed ≤ seven days before inclusion in the study)
* Recovery or stabilization to grade ≤ 1 from any adverse event derived from previous treatment (up to grade 2 alopecia or asthenia/fatigue are allowed).
* No clinically significant changes in ECG.
* At least four weeks since the last monoclonal antibody containing therapy or definitive radiotherapy (RT)
* At least two weeks since the last biological/investigational single-agent therapy (excluding MAbs) and/or palliative RT (≤10 fractions or ≤30 Gy total dose)
* Fertil women must have pregnancy excluded by appropriate testing before study entry

Exclusion Criteria:

* Prior treatment with PM01183 or trabectedin.
* Concomitant diseases/conditions:

  * History within the last year or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically relevant valvular heart disease or symptomatic arrhythmia or any asymptomatic ventricular arrhythmia requiring ongoing treatment.
  * Ongoing, non-neoplastic, chronically active liver disease of any origin.
  * Active infection.
  * Patients who are requiring any ongoing oxygen support.
  * Known human immunodeficiency virus (HIV) infection.
  * Any other major illness.
* Symptomatic or corticosteroid-requiring brain metastases or leptomeningeal disease involvement. Patients with asymptomatic documented stable brain metastases not requiring corticosteroids during the last three months are allowed.
* Peripheral sensory/motor neuropathy grade >1. Hearing impairment grade >1.
* Fertile men or women not using an effective method of contraception.
* History of bone marrow or stem cell transplantation
* Radiotherapye to >35% of the bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07-30; Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Recommended dose (RD) of the combination PM01183 and cisplatin | 30 months
  To determine the recommended dose (RD) of PM01183 in combination with cisplatin every three weeks (q3wk) with or without aprepitant in patients with advanced solid tumors. The RD will be the dose level (DL) immediately below the maximum tolerated dose (MTD), that is, the highest DL explored at which less than one third of evaluable patients experience a DLT during Cycle 1.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) characterisation of Cmax (maximum concentratio), AUC (area under the curve), CL (clearance), HL (half life) y Vss (volume of distribution) | 30 months
  To characterize the pharmacokinetics (PK) parameters Cmax (maximum concentratio), AUC (area under the curve), CL (clearance), HL (half life) y Vss (volume of distribution ) of this combination in patients receiving/not receiving aprepitant and to explore factors that may affect individual variability in main PK parameters.
Pharmacogenomic (PGx) analysis | 30 months
  To conduct an exploratory pharmacogenomic (PGx) analysis to identify and validate putative molecular markers associated with the clinical outcome of patients treated with PM01183 and cisplatin. These molecular markers would help in the future selection of patients who might preferentially benefit from PM01183 therapy, thus contributing to improve health care through a more individualized medicine.

CONTACTS AND LOCATIONS:
Locations (3):
- Bellinzona, Switzerland
- United Kingdom (2):
  - London
  - Newcastle

REFERENCES:
- [Derived] Metaxas Y, Kahatt C, Alfaro V, Fudio S, Zeaiter A, Plummer R, Sessa C, Von Moos R, Forster M, Stathis A. A phase I trial of lurbinectedin in combination with cisplatin in patients with advanced solid tumors. Invest New Drugs. 2022 Feb;40(1):91-98. doi: 10.1007/s10637-021-01142-1. Epub 2021 Aug 28. PMID 34453241